CLINICAL TRIAL: NCT03262623
Title: Localized Radial Nerve Block for Treatment of Tennis Elbow: a Prospective, Randomized Clinical Trial
Brief Title: Radial Nerve Block for Treatment of Tennis Elbow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Chairperson of Anesthesia and Pain Management Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1082017
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Pain, Elbow
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radial nerve block (Experimental): Patients will receive radial nerve block guided by a nerve stimulator.
  Interventions: Other: Radial nerve block
- Placebo (Placebo Comparator): Patients will receive placebo through radial nerve block
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Radial nerve block — A nerve stimulator will be used to localize the radial nerve. Then radial block will be performed. At this point 3-5 ml of the anesthetic mixture is injected. Each 10 ml of the anesthetic mixture contained: 3ml lidocaine 2%, 3ml lidocaine 2% with epinephrine, 1:2000,000, 3ml bupivicaine 0.5% and 1ml clonidine 150 µg/ml.
  Arms: Radial nerve block
Other: Placebo — A nerve stimulator will be used to localize the radial nerve. Then radial block will be performed containing normal saline
  Arms: Placebo

SUMMARY:
Background: Lateral epicondylitis, or tennis elbow, is a common musculoskeletal disorder that causes pain and functional limitation. Although different nonsurgical conservative therapies such as bracing, physical therapy, nonsteroidal anti-inflammatory drugs, and corticosteroid injections in addition to surgical approaches have been used, yet there is no standard treatment for lateral epicondylitis.

Objectives: The primary objective of this study is to assess the effectiveness of nerve stimulator guided radial nerve block for treatment of lateral epicondylitis. The primary outcome measure is pain measured through the Visual Analogue Scale (VAS) at 1 and 2 weeks.

Methods: This is a prospective randomized, double blind clinical trial. Patients will be randomly allocated into two groups. Group I will receive radial nerve block guided by a nerve stimulator. Group II patients will receive placebo through radial nerve block. Patients will be followed up for 2 weeks.

DETAILED DESCRIPTION:
Lateral epicondylitis, or tennis elbow, is a common musculoskeletal disorder that causes pain and functional limitation. It is a major arm disorder which occurs commonly in adults between 30 and 50 years, with an estimated prevalence of 1% to 3% in the general population. Lateral epicondylitis results from the overuse of the extensor muscles, causing inflammation or irritation of the tendon insertion. It is common in workers whose job requires manual and repetitive work .

Although different nonsurgical conservative therapies such as bracing, physical therapy, nonsteroidal anti-inflammatory drugs, and corticosteroid injections in addition to surgical approaches have been used, yet there is no standard treatment for lateral epicondylitis.

To our knowledge, there are no studies that used nerve-stimulator-guided radial nerve block for the treatment of lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* presenting with refractory elbow pain

Exclusion Criteria:

patients with:

* osteoarthritis,
* rheumatoid arthritis,
* olecranon bursitis,
* radial nerve entrapment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Pain score | 2 weeks
  Pain will be measured through the Visual Analogue Scale (VAS). The scale ranges between 0 and 10, with 0 being no pain and 10 maximum possible pain

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Naja, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon